CLINICAL TRIAL: NCT01828294
Title: Subcutaneous Ig Maintenance Therapy for Myasthenia Gravis
Acronym: SIMM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped by sponsor due to difficulty enrolling at site
Sponsor: St. Louis University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Ghazala Hayat, Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17005
Record Dates: First submitted 2011-11-01; First posted 2013-04-10 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Myasthenia Gravis
Keywords: MG
MeSH Terms: conditions — Myasthenia Gravis | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Population (Other): Study population will include patients (18-80 years old) with non-thymomatous myasthenia gravis MGFA Class II-IV receiving a minimum of 30mg of Prednisone daily and no other immunosuppression and no more 240 mgs per day of Cholinesterase inhibitor. Patients will receive Subcutaneous immunoglobulins weekly for 6 months.
  Interventions: Drug: Subcutaneous immunoglobulins

INTERVENTIONS:
Drug: Subcutaneous immunoglobulins — Immunoglobulins used subcutaneously for maintenance of other immune mediated disorders.
  Other Names: Hizentra

SUMMARY:
The study is being done with patients with Myasthenia Gravis (MG), age 18-80 years, positive acetylcholine receptor antibody, receiving greater than 30mg of prednisone daily. Patients may or may not be receiving anticholinesterase agents. A common treatment for patients with this disease includes the administration of intravenous immunoglobulin (IVIG), which is a plasma protein that is given to help maintain adequate antibody levels to prevent infections and decrease the symptoms of the disease of Myasthenia Gravis. This study is being done to test if giving this medication in a subcutaneous form (into the fat of the abdomen, legs and thighs) will be better tolerated for patients with Myasthenia Gravis.

DETAILED DESCRIPTION:
The study is a pilot study to ascertain the feasibility and tolerability of subcutaneous immunoglobulin (SCIG or IGSC) as a maintenance therapy for patients with non-thymomatous MG patients (MGFA class II-IV) at entry, aged 18-80 years, positive acetylcholine receptor antibody, receiving greater than 30mg of prednisone daily. Patients may or may not be receiving anticholinesterase agents.

The neurologist principal investigator at each site will have the overall responsibility for study performance is designated the medical coordinator (MC). The MC will assess patients from the sites clinic populations and identify potential subjects for inclusion and exclusion criteria. Once a subject is identified and provided informed consent to participate the Visit Schedule will be initiated.

At the initial visit the MC will perform the acetylcholine receptor antibody level, and record the prednisone and anticholinesterase doses. The MC will be responsible for assessment of adverse events. The research coordinator will arrange for the initial laboratory testing at the patient's local Quest, where the blood will be drawn. Baseline lab tests to be done will include IgA level to evaluate for deficiency, IgG level, CBC, AchR antibody, pregnancy tests in women, LFT's, PT/PTT and BUN/Creatinine. The patient will complete the SF-36 quality of life, MG, and MGFA ADL The research coordinator will be responsible for training subjects in performance of IGSC infusion. Subjects will have outpatient clinic assessments in one week and then monthly for the remainder of the study. Patients will receive 2gms/kg divided over 4 weeks initially and then will be given 250mgs/kg/wk for total of 6 months. This is similar to the standard IV treatment for patients which is 2 gm/kg given over 2-5 days for the initial dose. After the initial dose, a patient is started on monthly IV maintenance dose of 1 gm/kg each month given over 1-3 days.

The subject will be evaluated monthly for assessment of whether minimal manifestation (MM) status has been reached, which then allows reduction of corticosteroids by 5mg or more if clinically indicated. The MC will record adverse events and symptoms. The dose of anticholinesterase drugs will be decreased at the discretion of the MC. The prednisone dose will be decreased unless the MM status is lost; in that situation the prednisone dose will be increased 10mg every 2 weeks until the MM is again achieved. Titration of the prednisone and cholinesterase inhibitor medications will be at the discretion of the physician and will be based on the patient's symptoms as measured by symptoms and examination, leading to a determination of the MM. The patient will complete the SF-36 quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

1. AChR Ab positive myasthenia gravis (acetylcholine receptor antibody).
2. Age 18-80 years.
3. MGFA Classification II-IV (The scale used to determine the severity of symptoms of MG).
4. Receiving > or equal 30mg of Prednisone per day.
5. No new MG-specific treatments in prior 3 months.
6. Willingness to participate in study protocol.
7. QMG > 10 (quantitative myasthenia gravis score: the sum of grades given for symptoms of MG).
8. Treatment with any immunomodulator > than or equal to 3 months prior to trial initiation.

Exclusion Criteria:

1. IgA deficiency (a major class of immunoglobulins found in serum and external body secretions such as saliva, tears, and sweat as well as in the gastrointestinal, respiratory, and genitourinary tracts).
2. Previous thromboembolic events, including deep vein thrombosis, stroke and myocardial infarction
3. MGFA Class I, IV (if patient requires hospitalization) or V
4. History of thymoma
5. Thymectomy in previous year or planning to undergo thymectomy in next six months
6. Pregnancy or lactation; unwillingness to avoid pregnancy
7. Serious concurrent medical, neurological or psychiatric condition that would interfere with IGSC administration or subsequent clinical assessments
8. Unwillingness or incapacity to participate, agree to necessary follow-up visits, or give written and informed consent
9. Patients who have had an anaphylactic or severe systemic reaction to the administration of human immune globulin or to components of Hizentra, such as polysorbate 80, or patients with hyperprolinemia because it contains the stabilizer L-proline
10. Cholinesterase inhibitor no more than 240 mg/day
11. Body weight greater than 120 kg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To monitor number of participants completing the study for the six months period | Baseline to 6 months
  To evaluate feasibility and tolerability of IGSC as a maintenance treatment of generalized MG as measured by treatment adherence and adverse events experienced by the patient. Patients will be asked if they have experienced any of the most commonly known side effects of Hizentra. A case report form detailing any adverse events will be included with every study visit and reviewed with the patient at each visit.

SECONDARY OUTCOMES:
To monitor number of adverse events in participants | Baseline to 6 months
  •To evaluate safety IGSC for treatment of generalized MG as measured by adverse events experienced by each patient and reviewed monthly by the principal investigator.
Number of participants able to decrease prednisone dose below 30 mgs | Baseline to 6 months
  • To evaluate the potential steroid-sparing effect of IGSC treatment as measured by the total dose of prednisone required by each patient over the six month period.
To monitor effect on manual muscle testing | Baseline to 6 months
  • To evaluate the effect of IGSC treatment on symptoms associated with MG as measured by the QMG and MG-ADL.
To measure changes on SF-36 quality of life measurement tool before and after completion of study | Baseline to 6 months
  • To evaluate Quality of Life with IGSC treatment for MG as measured by the SF-36.
To measure and correlate levels of serum IgG with clinical response of the participants | Baseline to 6 months
  • To evaluate pharmacokinetics (IgG) levels associated with IGSC treatment for MG as measured by the monthly blood draws.
To monitor minimal manifestation of Myasthenia Gravis | Baseline to 6 months
  To evaluate the effect of IGSC treatment on symptoms associated with MG
To monitor effect on Quantitative Myasthenia Gravis Score | Baseline to 6 months
  To evaluate the effect of IGSC treatment on the Quantitative Myasthenia Score. Data collected will be qualitative and quantitative, and scores will be compared over time. Data will be captured on case report forms, and entered into an SPSS database. Dr. Gary Cutter, who is serving as a statistician for this study, will review the data monthly for safety, and a report will be sent to Dr. Hayat.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazala Hayat, M.D., Principal Investigator — St. Louis University; Jafar Kafaie, M.D., Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - Saint Louis University, St Louis, Missouri